CLINICAL TRIAL: NCT05426876
Title: The Effect of Competition Season on Shoulder Periarticular Structures, Muscle Strength, Range of Motion, Scapular Muscle Endurance and Upper Extremity Performance in Young Swimmers
Brief Title: The Effect of Competition Season on Physical Characteristic and Shoulder Periarticular Structures in Swimmers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aykut OZCADIRCI, Principal Investigator, Hacettepe University
Other Study IDs: GO21/1341
Record Dates: First submitted 2022-06-09; First posted 2022-06-22 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Image; Athletic Injuries; Upper Extremity
Keywords: ultrasonography; upper extremity; subacromial space; young swimmers; muscle strength; range of motion
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the effect of a competition season on shoulder periarticular structures, muscle strength, muscle endurance, joint range of motion and upper extremity performance in young swimmers.

DETAILED DESCRIPTION:
After being informed about the study, all swimmers giving written informed consent will undergo a 1- week screening period to determine eligibility for study entry. Swimmers who meet the eligibility requirements will be evaluated 3 times: pre-season, mid-season, and post-season.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 10-15
* At least 6 hours of swimming training per week,
* Individuals do not have cooperation and communication problems,
* Individuals volunteer to participate in the study.

Exclusion Criteria:

* Previous upper extremity surgery,
* Experienced upper extremity pain at least 2 times in the past,
* Not attending training regularly for any reason.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In this study, volunteer swimmers who practice swimming professionally in Ankara University Sports Club will be evaluated and included in the study. In determining the sample size of the study, Tate et al. Data showing the difference in shoulder joint range of motion were used. As a result of the power analysis, it was determined that 23 participants should be included in such a way that the type 1 error was 5% and the power of the study was at least 95%. Considering the possibility of participants leaving the study during the study period, 30 swimmers were planned to be included in the study. Posthoc power analysis will be done with the data to be obtained after the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Changes in shoulder periarticular structures during training season | up to 32 weeks
  Measurements will be made by a medical physician with at least 4 years of experience in musculoskeletal ultrasonography. The participants will be placed in a position called the Crass position, where the arm is in extension, adduction, and internal rotation, and the dorsal aspect of the hand is placed on the lumbar region.
  Deltoid muscle thickness: The thickness of the muscle tissue between the skin and subcutaneous tissue and the supraspinatus tendon will be measured from the point where it is thickest.
  Supraspinatus tendon thickness: The supraspinatus muscle, which is between the deltoid muscle and the humerus-articular cartilage, will be measured at its thickest point.
  Cartilage thickness of the humeral head: Articular cartilage thickness, which is seen anechoic between the humerus and the supraspinatus tendon, will be measured from the midpoint.
  Acromiohumeral distance: The distance between the humerus and acromion will be measured in the neutral position.
Changes in muscle strength during the training season | up to 32 weeks
  Isometric muscle strength will be measured with a hand dynamometer. Before starting the measurement, the participants will be informed verbally about the technique of practice of the test. In order to ensure correct movement, individuals will be asked to perform a submaximal contraction against the evaluator's hand before the test and the measurements will be taught. The "break test" technique, which requires isometric contraction, will be applied during the tests. During the break test, the person performing the test pushes the dynamometer towards the patient's extremity until the movement is released in the relevant joint in a way that can overcome the maximum muscle strength.
  Bilateral shoulder flexion, extension, internal rotation, and external rotation muscle strength and serratus anterior, middle, and lower trapezius will be measured and averaged in 3 repetitions and recorded in "kg". A 30-second rest will be given between measurements.
Changes in Shoulder Range of Motion during training season | up to 32 weeks
  Both shoulder joint flexion, extension, internal and external rotation normal joint movements will be measured and recorded in degrees with a digital goniometer.
Changes in Upper Extremity Functional Performance during training season | up to 32 weeks
  The closed kinetic chain upper extremity stabilization test, which is a dynamic test, is used to evaluate potential strength and muscular strength deficits, as well as proprioception and motor control. The test is performed in a modified push-up position with elbows straight and knees bent. When the test is started, they will be asked to raise one of their hands and touch the other hand, and the number of times the athletes touched their hands within 15 seconds will be recorded.
Assessment of Scapular Muscle Endurance | up to 32 weeks
  Muscle endurance will be assessed using the posterior shoulder endurance test. While the measurement is lying prone, participants will be asked to actively raise their arms to a horizontal position at an angle of 135 ('Y' position). A movable clamp to be placed on a vertically oriented metal bar will be set to mark the point where the radial direction of the wrist contacts the horizontal bar. The swimmer will then lift a dumbbell of 1.0 or 1.5 kg (2% of body weight) and hold it at the final point and the holding time will be recorded with the stopwatch. The test will begin when the swimmer's wrist is in contact with the clamp and will be terminated if compensation occurs, such as loss of arm contact with the bar or trunk rotation.

SECONDARY OUTCOMES:
Anthropometric measurements | at baseline
  Participants' height in cm will be measured. In addition, parameters such as arm span, shoulder width, arm length, and sitting and standing height will be measured in cm and recorded.
Body weight measurement | at baseline
  The body weight of the participants will be measured and recorded in kilograms.
Body Mass Index | at baseline
  Body mass index is obtained by dividing the body weight in kilograms by the square of the height in meters. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Body Composition measurement | at baseline
  Body composition will be evaluated with a bioelectrical impedance analyzer (BIA) device InBody 120 (IB120) (InBody USA) with tetrapolar-8 point tactile electrodes. The participants will step on the scale with bare feet and light clothes, aligning their heels and feet with the electrodes on the measuring scale, to ensure maximum contact area, and they will be asked to stand still while their body mass is measured. To ensure that the arms do not touch the trunk during the measurement, the participants will be positioned with the elbows in full extension and the arms in approximately. The device has two frequencies (20 and 100 kHz) for impedance measurement in five body segments (four extremities and trunk). Body composition parameters used; total body muscle mass (SMM; in kg), the lean mass of five body segments (FFM; in kg) and total body fat mass (BFM; in kg), and fat mass of five body segments.

IPD SHARING:
Plan to Share IPD: No